CLINICAL TRIAL: NCT05126888
Title: A Randomized, Double-Blind, Placebo Controlled, Cross-Over Study to Evaluate the Efficacy, Safety and Tolerability of Daily Oral SCI-110 in Treating Adults With Tourette Syndrome.
Brief Title: SCI-110 in the Treatment of Tourette Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurothera Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCI-021-001
Record Dates: First submitted 2021-10-25; First posted 2021-11-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SCI-110 (Experimental): Cannabinoid-based medication consisting of Dronabinol and PEA
  Interventions: Drug: SCI-110
- Dronabinol (Placebo Comparator): Placebo matched in taste, odour and appearance to SCI-110
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SCI-110 — SCI-110 - a softgel capsule containing Dronabinol and Palmitoylethanolamide (PEA) in the following doses: 2.5mg Dronabinol+400mg PEA, 5mg Dronabinol+400mg PEA and 10mg Dronabinol+400mg. Maximum dose 20mg Dronabinol and 800mg PEA a day.
  Arms: SCI-110
Other: Placebo — Pill that matches in taste, odour and appearance to SCI-110 active pills
  Arms: Dronabinol

SUMMARY:
To evaluate the efficacy, safety and tolerability of the cannabinoid-based medication SCI-110 compared to placebo in subjects with Tourette syndrome.

DETAILED DESCRIPTION:
It is believed that SCI-110 will be a valuable treatment option, especially for t those subjects with TS, who do not benefit from or do not tolerate first-line treatment with antipsychotics. Since there is evidence that currently available CBM improves not only tics, but also psychiatric comorbidities, SCI-110 might be even more beneficial to improve a broader spectrum of symptoms resulting in both improved quality of life and decreased disease related costs. Moreover, PEA was shown to minimize AEs associated with cannabinoids use and to reduce their required effective dose (data not published). Hence, the use of SCI-110 is expected to show a therapeutic effect superior to currently available CBMs.

It can be assumed that AEs in TS subjects do not differ from AEs described in other groups of subjects treated with medicinal cannabis and/or cannabinoids. In general, cannabinoids are considered as well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Tourette syndrome according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
2. Male and female subjects with an age between ≥18 and ≤65 years
3. Total tic score (TTS) of the revised Yale Global Tic Severity Scale (YGTSS-R) >14
4. Clinical Global Impression-Severity Score (CGI-S) ≥4
5. Medication (and stimulation parameters for deep brain stimulation) for tics and comorbidities must be on a stable dose for at least 6 weeks before entering the study and subject must consent to maintain the stable dose during the study
6. Signed written informed consent and willingness to comply with treatment and follow-up procedures
7. Subjects capable of understanding the investigational nature, potential risks and benefits of the clinical study
8. Women of child-bearing potential must have a negative pregnancy test (e.g., urine human chorionic gonadotropin [hCG]) before first treatment with study medication. They must practice a highly effective, reliable and medically approved contraceptive regimen during the study (e.g., theoretical failure rate less than 1% per year as when used consistently and correctly), which include oral or parenteral or implanted hormonal contraception, vaginal ring releasing hormonal contraception (e.g., Nuvaring), intrauterine device or intrauterine system. Women without childbearing potential may enter this study. Women without childbearing potential defined as follows:

   * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
   * hysterectomy or uterine agenesis or
   * ≥ 50 years and in postmenopausal state ≥ 1 year or
   * < 50 years and in postmenopausal state ≥ 1 year with urine FSH > 40 IU/l and urine oestrogen < 30 ng/l, or serum follicle stimulating hormone (FSH) in the post-menopausal range or a negative oestrogen test.
9. Male subjects must be willing to use a condom with sexual partners during this study and for a period of three months following the last administration of study medication until the follow-up visit. Male subjects must be willing to abstain from sperm donation for 3 months after the completion of this study

Exclusion Criteria:

1. Comorbid obsessive-compulsive disorder (OCD), attention deficit/hyperactivity disorder (ADHD), depression, and anxiety disorder when unstable or in need of an initial adjustment for a therapy-according to the investigator's judgment
2. Presence of severe psychiatric conditions such as developmental disability, psychotic illness and bipolar disorder- according to the investigator's judgment
3. Ongoing behavioural treatment for tics
4. History of schizophrenia, seizure, psychotic, severe personality, or pervasive developmental disorder
5. Current clinical diagnosis of substance abuse or dependence
6. History of cannabis dependence
7. Secondary and other chronic tic disorders or other significant neurological disorders
8. Known severe cardiac diseases, known severe cardiovascular diseases, known positivity for human immunodeficiency virus (HIV), hepatitis C, hepatitis B, or other severe hepatic and renal disorders by history
9. Concomitant medications have to be on stable dose since at least 6 weeks before entering the study and must be well tolerated at baseline without causing dizziness, confusion, sedation, or somnolence)
10. Use of cannabis or cannabinoid-based medicine (CBM) in the 30-day period prior to study entry and/or positive delta-9-tetrahydrocannabinol (THC) urine test at baseline
11. Positive urine ß-HCG pregnancy test
12. Pregnant or breast-feeding women
13. Subjects who received any investigational medication or used any investigational device within 30 days prior to the first dose of study medication or is actively participating in any investigational drug or device study, or is scheduled to receive an investigational drug or to use an investigational device during the course of the study
14. Subjects with a known allergy, hypersensitivity, or intolerance to the active substances and ingredients of study medication (e.g., cannabis, cannabinoids, or sesame oil)
15. Any condition, which in the opinion of the investigator, would interfere with the evaluation of the study product or poses a health risk to the subject
16. Subjects who are employees of the sponsor or employees or close relatives of the investigator
17. Subjects with active suicidal ideation and behaviour (SI/B) according to the Columbia-Suicide Severity Rating Scale (C-SSRS) and/or subjects that have attempted suicide in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in revised version of Yale Global Tic Severity Scale -Revised - (YGTSS-R-TTS) | At baseline and 12 weeks after start of treatment in both arms.
  Absolute change from baseline in revised version of YGTSS-R-TTS as a continuous endpoint at week 12 of the respective treatment period.
  The Global Severity Score has a range of 0- 100. A higher score on the scale suggests a more severe Tic, or a greater impact the Tic has on the person's life.

SECONDARY OUTCOMES:
Percent reduction in Yale Global Tic Severity Scale -Revised - (YGTSS-R-TTS) of at least 20% | At baseline and 12 weeks after start of treatment in both arms.
  Response to treatment according to YGTSS-R-TTS of at least 20% reduction (compared to baseline)
  The responder criterion defined as a more severe Tic, or a greater impact the Tic has on the person's life The Global Severity Score has a range of 0- 100. A higher score the scale suggests a more severe Tic, or a greater impact the Tic has on the person's life.
Percent reduction in Yale Global Tic Severity Scale -Revised - (YGTSS-R-TTS) of at least 30%, 35% and 50% | Week 12 of each treatment period (visit 8 and 15).
  Response to treatment according to YGTSS-R-TTS responder criterion, defined as a percent reduction in YGTSS-R-TTS of at least 30%, 35% and 50% (compared to baseline) The Global Severity Score has a range of 0- 100. A higher score on the scale suggests a more severe Tic, or a greater impact the Tic has on the person's life.
Absolute change from baseline of YGTSS-R Total Score | At baseline and 12 weeks after start of treatment in both arms.
  Absolute change from baseline of YGTSS-R Total Score, the corresponding subdomain motor and phonic total tic scores, the YGTSS-R Impairment Score, as well as of the combination of the total tic score and the impairment score (YGTSS-R-GS (= YGTSS-R-TTS + YGTSS-R-impairment score).
Percent change from baseline of YGTSS-R Total Score | At baseline and 12 weeks after start of treatment in both arms.
  Percent change from baseline of YGTSS-R Total Score, the corresponding subdomain motor and phonic total tic scores, the YGTSS-R Impairment Score, as well as of the combination of the total tic score and the impairment score (YGTSS-R-GS (= YGTSS-R-TTS + YGTSS-R-impairment score).
Clinical Global Impression-Improvement Score (CGI-I) | 24 weeks
  Absolute values of the Clinical Global Impression-Improvement Score (CGI-I). CGI is a 7 point scale that ranges from 1 Very much improved to 7 Very much worse
Clinical Global Impression-Severity Score (CGI-S) Absolute result | 24 weeks
  Absolute change from baseline of Clinical Global Impression-Severity Score (CGI-S).
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  The range is from 1 Normal, not at all ill to 7 Among the most extremely ill patients
Clinical Global Impression-Severity Score (CGI-S) Percent result | 24 weeks
  Percent change from baseline of Clinical Global Impression-Severity Score (CGI-S).
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  The range is from 1 Normal, not at all ill to 7 Among the most extremely ill patients
Total Pre-monitory Urge for Tics Scale (PUTS) Absolute Score | 24 weeks
  Absolute change from baseline of the total Pre-monitory Urge for Tics Scale (PUTS) Score.
  The range of the test is between 9 - 36. A higher score on the scale indicates an extremely high intensity with probable severe impairment.
Total Pre-monitory Urge for Tics Scale (PUTS) Percent Score | 24 weeks
  Percent change from baseline of the total Pre-monitory Urge for Tics Scale (PUTS) Score.
  The range of the test is between 9 - 36. A higher score on the scale indicates an extremely high intensity with probable severe impairment.
Adult Tic Questionnaire (ATQ) Percent Score | 24 weeks
  Percent change from baseline of the total Adult Tic Questionnaire (ATQ) Score. The Adult Tic Questionnaire (ATQ) Score has a range of 0- 50. A higher score on all scales suggests a more severe Tic, or a greater impact the Tic has on the person's life.
Adult Tic Questionnaire (ATQ) Absolute Score | 24 weeks
  The absolute change from baseline of the total Adult Tic Questionnaire (ATQ) Score.
  The Adult Tic Questionnaire (ATQ) Score has a range of 0- 50. A higher score on all scales suggests a more severe Tic, or a greater impact the Tic has on the person's life.
Changes in Beck Depression Inventory (BDI-II) Percent score. | 24 weeks
  Percent change from baseline of the Beck Depression Inventory (BDI-II) total score The questionnaire contains about 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression
Changes in Beck Depression Inventory (BDI-II) absolute score. | 24 weeks
  Absolute change from baseline of the Beck Depression Inventory (BDI-II) total score The questionnaire contains about 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression
Changes in Yale-Brown Obsessive Compulsive Scale (Y BOCS) absolute score | 24 weeks
  Absolute change from baseline of the Yale-Brown Obsessive Compulsive Scale (Y BOCS) Total scores on the measure range from 0 to 40, with a score of 0-7 indicating subclinical symptoms, 8-15 mild symptoms, 16-23 moderate symptoms, 24-31 severe symptoms and 32-40 extreme symptoms.
Changes in Yale-Brown Obsessive Compulsive Scale (Y BOCS) Percent score | 24 weeks
  Percent change from baseline of the Yale-Brown Obsessive Compulsive Scale (Y BOCS) score.
  Total scores on the measure range from 0 to 40, with a score of 0-7 indicating subclinical symptoms, 8-15 mild symptoms, 16-23 moderate symptoms, 24-31 severe symptoms and 32-40 extreme symptoms.
Changes in Obsessive-compulsive disorder (OCD) severity Absolute score | 24 weeks
  Absolute change from baseline of the total Obsessive-compulsive disorder (OCD) severity score.
  The range of the test is between 8-15 = Mild OCD; 16-23 = Moderate OCD; 24-31= Severe OCD; 32-40 = Extreme OCD
Changes in Obsessive-compulsive disorder (OCD) severity Percent score | 24 weeks
  Percent change from baseline of the total Obsessive-compulsive disorder (OCD) severity score.
  The range of the test is between 8-15 = Mild OCD; 16-23 = Moderate OCD; 24-31= Severe OCD; 32-40 = Extreme OCD
Changes in Conners' Adult ADHD Rating Scale (CAARS) Absolute score. | 24 weeks
  Absolute change from baseline of the Conners' Adult ADHD Rating Scale (CAARS) score.
  When total score is less than 60 there is no indication of ADHD. A score higher than 60 may indicate ADHD. And a total score higher than 70 means ADHD with more serious symptoms.
Changes in Conners' Adult ADHD Rating Scale (CAARS) Percent score | 24 weeks
  Percent change from baseline of the Conners' Adult ADHD Rating Scale (CAARS) score When total score is less than 60 there is no indication of ADHD. A score higher than 60 may indicate ADHD. And a total score higher than 70 means ADHD with more serious symptoms.
Changes in Beck Anxiety Inventory (BAI) Absolute scores | 24 weeks
  Absolute and percent change from baseline of the Beck Anxiety Inventory (BAI) The BAI assessments contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are: 0-7: Minimal, 8-15: Mild, 16-25: Moderate and 26-63: Severe
Changes in Beck Anxiety Inventory (BAI) percent scores | 24 weeks
  Percent change from baseline of the Beck Anxiety Inventory (BAI) score. The BAI assessments contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are: 0-7: Minimal, 8-15: Mild, 16-25: Moderate and 26-63: Severe
Changes in Beck Depression Inventory (BDI) Absolute score | 24 weeks
  Absolute change from baseline of the total BDI score. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows: 0-9: indicates minimal depression, 10-18: indicates mild depression, 19-29: indicates moderate depression, 30-63: indicates severe depression. Higher total scores indicate more severe depression
Changes in Beck Depression Inventory (BDI) percent score | 24 weeks
  Percent change from baseline of the total BDI score. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows: 0-9: indicates minimal depression, 10-18: indicates mild depression, 19-29: indicates moderate depression, 30-63: indicates severe depression. Higher total scores indicate more severe depression
Changes in Rage Attacks Questionnaire (RAQ-R) Absolute scores | 24 weeks
  Absolute change from baseline of the Rage Attacks Questionnaire (RAQ-R) score. The RAQ-R assessments contains 22 questions, each answer being scored on a scale value of 0 (not at all) to 4 (Very powerful, very common). Higher total scores indicate more severe Rage Attacks.
Changes in Rage Attacks Questionnaire (RAQ-R) percent scores | 24 weeks
  Percent change from baseline of the Rage Attacks Questionnaire (RAQ-R) score. The RAQ-R assessments contains 22 questions, each answer being scored on a scale value of 0 (not at all) to 4 (Very powerful, very common). Higher total scores indicate more severe Rage Attacks.
Changes in Pittsburgh Sleep Quality Index (PSQI) Absolute scores | 24 weeks
  Absolute change from baseline of the Pittsburgh Sleep Quality Index (PSQI) global score.
  PSQI Consisting of 19 items, Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Changes in Pittsburgh Sleep Quality Index (PSQI) Percent scores | 24 weeks
  Percent change from baseline of the Pittsburgh Sleep Quality Index (PSQI) global score.
  PSQI Consisting of 19 items, Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Changes to the Tourette Syndrome-Quality of Life Scale (GTS-QoL) score | 24 weeks
  Changes from baseline of Tourette Syndrome-Quality of Life Scale (GTS-QoL). GTS-QoL is a 27-item, self-report questionnaire that assesses HR-QoL in young patients with tic disorders, encompassing 4 areas of HR-QoL: psychological, physical/activities of daily living, obsessive-compulsive, and cognitive domains. Each item is rated on a 5-point Likert-type scale and higher scores indicate worse HR-QoL. The instrument includes a Visual Analogue Scale used to express the extent of self-satisfaction about life (higher scores indicate higher satisfaction)
Changes to the 12-item short-form Health Survey (SF-12) score | 24 weeks
  Changes from baseline of 12-item short-form Health Survey (SF-12). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

OTHER OUTCOMES:
Number and rate of patients affected by AEs, SAEs, SUSARs/ADRs, AESIs and AEs | 24 weeks
  Number of adverse events (AEs), number and rate of patients affected by AEs, Serious Adverse Events (SAE), Suspected Unexpected Serious Adverse reactions (SUSAR) /Adverse Drug Reaction (ADR), Adverse Events of Special Interest (AESI) and AEs leading to withdrawal at each visit.
Absolute values of vital sign blood pressure at each visit and change from baseline. | 24 weeks
  Absolute values of vital sign blood pressure at each visit and change from baseline for each visit. Number and percentage of clinically significant abnormal values.
Absolute values of vital sign heart rate at each visit and change from baseline. | 24 weeks
  Absolute values of vital sign heart rate at each visit and change from baseline for each visit. Number and percentage of clinically significant abnormal values.
2.3. Suicide risk assessment measured by the Columbia-Suicide Severity Rating Scale (CSSRS) | Through out the study
  Suicide risk assessment measured by the Columbia-Suicide Severity Rating Scale (CSSRS) and change from baseline for each on-site visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten R Müller-Vahl, PhD. MD, Principal Investigator — Hannover Medical School
Locations (3):
- Yale Child Study Center - NIHB 205, New Haven, Connecticut, United States
- Medizinische Hochschule Hannover, Hanover, Germany
- Neurological Institute, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No